CLINICAL TRIAL: NCT05800652
Title: The Effect of the Peer Mentoring Program Applied to Nursing Students on Perceived Stress and Self-confidence
Brief Title: Mentoring Program for Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Merve Kızılırmak Tatu, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MTatu
Record Dates: First submitted 2023-03-24; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Mentoring; Nursing Students
Keywords: peer mentoring; self-efficacy; self-confidence; perceived stress; nursing students

STUDY DESIGN:
Intervention Model Description: Study has been planned as a type of randomized controlled intervention type with pre -test and monitoring patterns, one of the quantitative research methods. 40 mentees/first year students (experimental = 20; control = 20) and 20 mentors/fourth year students were included in the study. Simple random randomization was used in the appointment of the students in the sample group to experimental and control groups. Mentors were randomly matched with the mentees assigned to the experimental group.12 -week mentoring program was applied to the mentees by the mentors. In the collection of research data, "Personal Information Form", "General Self -Qualification Scale", "Self -Confidence Scale" and "Perceived Stress Scale" were used. The measurements were taken 3 times:pre test, post-test and 3-months post-test.
Who Masked: Participant, Outcomes Assessor
Masking Description: In this study, the analysis of the data was conducted by an independent statistician who does not know the intervention and control group appointment. In addition, students were not explained in which group they were in and they were blinded.Simple random randomization was used in the appointment of the students in the sample group to experimental and control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Experimental: First-year nursing students (mentees) undergoing a mentoring program 20 mentees were included in the experimental group.The mentoring program focuses on developing students' life skills. The mentoring program continued for 12 weeks. In the mentoring program, it was expected that the mentors would make individual meeting(s) with the mentee they were matched with, face to face, online or over the phone, and share information and support every week. The frequency and duration of individual interviews were determined by the needs of the mentee.
  Interventions: Behavioral: Peer Mentoring Program
- Control (No Intervention): No Intervention: Control group 20 mentees were included in the control group. After the follow-up test was applied to the students in the experimental group, a three-week mentoring program was applied to the control group.

INTERVENTIONS:
Behavioral: Peer Mentoring Program — Mentoring program created in academic, social, emotional and safety dimensions.In the academic dimension, there is information about the instructors, course selection, preparing a course study program,efficient study methods,information about the education and training program. Social dimension includes interpersonal relations, participation in social life, free time activities, making friends.The emotional dimension includes developing self-confidence,coping with stress,belonging and motivation.In the security dimension, there are student rights,scholarship opportunities, accommodation opportunities, library and internet facilities, use of the health center and clinical practice. In the mentoring program, it was expected that the mentors would make individual meeting(s) with the mentee they were matched with, face to face, online or over the phone, and share information and support every week. The mentoring program continued for 12 weeks.
  Arms: Experimental

SUMMARY:
University life is a challenging period for many students. University students mostly leave their families and live in crowded environments such as home and home. Research shows that students have difficulty in adapting to university life and often experience emotional, academic, professional and economic problems. Peer mentoring is one of the methods of learning and developing life skills in meeting the needs of university students.The peer mentoring intervention, which is used effectively in nursing education, provides benefits to both mentor and menene; It provides the opportunity to grow and improve by improving positive interaction between peers.It can be said that peer mentoring has a significant effect on students in line with the literature information. In this study, it was planned to examine the impact of the peer mentoring program applied on the perceived stress and self -confidence in order to ensure that the first year students of the nursing students adapt to the university life and the profession and to gain the necessary skills to survive in this process.

DETAILED DESCRIPTION:
In this study, it was planned to examine the impact of the peer mentoring program applied on the perceived stress and self -confidence in order to ensure that the first year students of the nursing students adapt to the university life and the profession and to gain the necessary skills to survive in this process. Study has been planned as a type of randomized controlled intervention type with pre -test and monitoring patterns, one of the quantitative research methods. 40 mentees (experiment = 20; control = 20) and 20 mentors were included in the study.12 -week mentoring program was applied to the mentees by the mentors. In the collection of research data, "Personal Information Form", "General Self -Qualification Scale", "Self -Confidence Scale" and "Perceived Stress Scale" were used. The measurements were taken 3 times:pre test, post-test and 3-months post-test.

ELIGIBILITY:
Inclusion Criteria:

* volunteering to participate in the study

Exclusion Criteria:

* being a foreign national
* taking first-year courses repeatedly
* be in another ongoing mentoring or psychosocial support/counselling program

Ages: 17 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
General Self-Efficacy Scale (GSE) | Change from baseline to 12 weeks (also assessed at 24 weeks post-baseline)
  The scale aims to determine the general self-efficacy level of individuals. The scale has 10 items and one dimension, and has a 4-point Likert (1=completely false- 4=completely true=) structure. The score obtained from the scale is between 10-40. A high score means high general self-efficacy.
Perceived Stress Scale (PSS) | Change from baseline to 12 weeks (also assessed at 24 weeks post-baseline)
  The scale, which consists of a total of 14 items, was designed to measure how stressful some situations in the life of the individual are perceived. The scale is 5-point Likert type. A score between 0 and 56 is taken from the scale. A high score indicates an excess of one's perception of stress.
Self-Confidence Scale (SCS) | Change from baseline to 12 weeks (also assessed at 24 weeks post-baseline)
  The scale consists of 33 items and 2 subscale. The scale is arranged in a 5-point Likert style and the maximum score that can be obtained from the scale is 165. A high score from the scale without reverse coded items indicates a high level of self-confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Kızılırmak Tatu, Principal Investigator — Gazi University Nursing Faculty, Ankara, Turkey
Locations (1):
- Merve Kızılırmak Tatu, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Other researchers will be able to read detailed information such as the research method and results when the research is published. The "Research Protocol" will be available on the this PRS page.